CLINICAL TRIAL: NCT07015359
Title: Evaluation of the Effect of Spinal Anesthesia-Induced Hypotension on Renal Functions in Preeclamptic Pregnant Women Using Neutrophil Gelatinase-associated Lipocalin (NGAL) and Standard Renal Function Tests
Brief Title: Renal Functions in Preeclamptic Pregnant Women Using Neutrophil Gelatinase-associated Lipocalin (NGAL) and Standard Renal Function Tests
Status: Not yet recruiting | Type: Observational
Sponsor: Nihan Aydin Guzey (Other)
Collaborators: Ankara City Hospital Bilkent (Other)
Responsible Party: Sponsor-Investigator, Nihan Aydin Guzey, Assoc.Prof. MD, Ankara City Hospital Bilkent
Organization: Ankara City Hospital Bilkent (Other)
Other Study IDs: TABED 2/170/2024
Record Dates: First submitted 2025-05-26; First posted 2025-06-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Anesthesia; Spinal Aneshtesia; Acute Kidney Failure; Spinal Anesthesia Induced Hypotension; Preeclampsia (PE)
Keywords: Preeclampsia; Hypotension; NGAL; Creatinine; AKI
MeSH Terms: conditions — Acute Kidney Injury; Pre-Eclampsia; Hypotension

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CASE GROUP: During the operation, heart rate (HR) and peripheral oxygen saturation (SpO₂) were continuously monitored. Systolic arterial pressure (SAP), diastolic arterial pressure (DAP), and mean arterial pressure (MAP) were measured and recorded every 2 minutes for the first 15 minutes, then every 5 minutes thereafter. Hypotension was defined as a ≥30% decrease in MAP from baseline or systolic blood pressure <100 mmHg. Patients who developed hypotension within the first four measurements were included in the hypotension group. Patients who developed hypotension in later measurements were excluded from the study to avoid confusion with bleeding-related hypotension. A 5 mg bolus of ephedrine was administered to raise the MAP to 80% or more of the baseline level within 60 seconds. Surgical duration, amount of fluids administered, duration and number of hypotensive episodes, total dose of ephedrine, estimated blood loss, use of additional uterotonics or tranexamic acid, neonatal weight, and Apgar.
- CONTROL GROUP: During the operation, the patient's heart rate (HR) and peripheral oxygen saturation (SpO₂) were continuously monitored. Systolic arterial pressure (SAP), diastolic arterial pressure (DAP), and mean arterial pressure (MAP) were measured and recorded every 2 minutes for the first 15 minutes, and then every 5 minutes thereafter. Patients whose MAP did not decrease by 30% or more from the baseline value were considered the control group

SUMMARY:
Acute kidney injury (AKI) is a significant postoperative complication. Risk factors for AKI include impaired renal perfusion, decreased functional renal reserve, as well as advanced age, peripheral arterial disease, diabetes mellitus, renovascular disease and congestive heart failure. Mean arterial pressure (MAP) below 55-60 mmHg has been associated with postoperative AKI. Traditional diagnostic criteria for AKI include increased serum creatinine levels and oliguria. However, creatinine levels do not rise until more than half of renal function is lost. Serum and urine NGAL levels rise earlier-within 24-48 hours-making it a promising early biomarker.

In our study, hypotension is defined as systolic blood pressure <100 mmHg or a >30% decrease in MAP. Patients requiring ephedrine under these conditions will be evaluated as the hypotension group and compared with non-hypotensive patients in terms of NGAL, BUN (blood urea nitrogen), creatinine, and GFR (Glomerular Filtration Rate) values at baseline and at the 4th postoperative hour.

DETAILED DESCRIPTION:
All patients were informed about the study in the preoperative period and written informed consent was obtained before the procedure. The following data were recorded: age, sex, weight, height, BMI (Body Mass Index), comorbidities, regular medications, ASA (American Society of Anesthesiologists) classification, gestational age, history of preeclampsia in previous pregnancies, hemodynamic values and laboratory results. After being admitted to the cesarean operating room, patients were monitored according to the ASA guidelines using standard monitoring methods (non-invasive arterial blood pressure measurements at 2-minute intervals, 3-lead ECG (Electrocardiogram) and pulse oximetry). A peripheral intravenous line was established via the dorsum of the hand and Ringer's lactate was infused at a rate of 10 mL/kg/h. All patients received oxygen via nasal cannula at a rate of 3-4 L/min.

Blood samples were collected from the patients before spinal anesthesia and at the 4th postoperative hour. The samples were centrifuged at 4000×g for 10 minutes in the biochemistry laboratory and then transferred into Eppendorf tubes and stored at -80°C in a deep freezer until the day of analysis. NGAL levels were measured using an ELISA (Enzyme-Linked ImmunoSorbent Assay) method with a commercial kit (USCN, China) at the Biochemistry Laboratory of Ankara Bilkent City Hospital. Each sample was measured in duplicate, and the mean values were used for evaluation. The intra-assay and inter-assay coefficients of variation (CV%) for the kit were determined to be <10% and <12%, respectively. At the 4th postoperative hour, blood samples were also analyzed for BUN, creatinine, and GFR levels, which were recorded accordingly.

ELIGIBILITY:
Inclusion Criteria:

* Patients classified as ASA physical status II-III
* Pregnant women aged 18-45 years, diagnosed with preeclampsia and scheduled for elective cesarean section, will be included in the study.

Exclusion Criteria:

* Patients who are unable to read, understand, or sign the informed consent form
* Patients with a diagnosed renal disease
* Patients who do not wish to participate in the study
* Patients with ASA physical status greater than III
* Patients younger than 18 or older than 45 years
* Patients requiring sedation or undergoing general anesthesia
* Patients with cardiac instability
* Patients with known arrhythmias

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Preeclamptic pregnant women aged 18 to 45 years, classified as ASA II-III, who volunteered to participate, were scheduled for cesarean section, and received spinal anesthesia were included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 46 (Estimated)
Dates: Start 2025-06-08 (Estimated); Primary Completion 2025-09-22 (Estimated); Study Completion 2025-10-20 (Estimated)

PRIMARY OUTCOMES:
ID: TABED 2/170/2024 Change in Plasma NGAL Levels Before and After Spinal Anesthesia | Before spinal anesthesia and at postoperative 4th hour
  To assess whether spinal anesthesia-induced hypotension in preeclamptic patients leads to early kidney injury, based on changes in plasma NGAL (neutrophil gelatinase-associated lipocalin) levels.

SECONDARY OUTCOMES:
Renal Function Parameters Post-Spinal Anesthesia | Postoperative 4th hour
  Evaluation of postoperative serum urea levels to assess renal function in the early postoperative period.
Comparative Timing of NGAL and Creatinine in Detecting AKI | NGAL measured before and 4 hours after anesthesia; creatinine at 4 hours
  To compare the timing of elevation between plasma NGAL and serum creatinine for early detection of acute kidney injury in preeclamptic patients.
Intraoperative Hemodynamic Monitoring | Measurements recorded at 2, 4, 6, 8, 10, 12, 14, 20, 25, 30, 35, 40, 50, and 55 minutes after spinal anesthesia initiation.
  Measurement of hemodynamic parameter systolic arterial pressure [SAP] at specified time points during the operation to evaluate the cardiovascular effects of spinal anesthesia in preeclamptic patients.
Intraoperative Hemodynamic Monitoring | Measurements recorded at 2, 4, 6, 8, 10, 12, 14, 20, 25, 30, 35, 40, 50, and 55 minutes after spinal anesthesia initiation.
  Measurement of hemodynamic parameter diastolic arterial pressure [DAP] at specified time points during the operation to evaluate the cardiovascular effects of spinal anesthesia in preeclamptic patients.
Intraoperative Hemodynamic Monitoring | Measurements recorded at 2, 4, 6, 8, 10, 12, 14, 20, 25, 30, 35, 40, 50, and 55 minutes after spinal anesthesia initiation.
  Measurement of hemodynamic parameter mean arterial pressure [MAP] at specified time points during the operation to evaluate the cardiovascular effects of spinal anesthesia in preeclamptic patients.
Intraoperative Hemodynamic Monitoring | Measurements recorded at 2, 4, 6, 8, 10, 12, 14, 20, 25, 30, 35, 40, 50, and 55 minutes after spinal anesthesia initiation.
  Measurement of hemodynamic parameter heart rate [HR] at specified time points during the operation to evaluate the cardiovascular effects of spinal anesthesia in preeclamptic patients.
Intraoperative Hemodynamic Monitoring | Measurements recorded at 2, 4, 6, 8, 10, 12, 14, 20, 25, 30, 35, 40, 50, and 55 minutes after spinal anesthesia initiation.
  Measurement of hemodynamic parameter oxygen saturation [SpO₂] at specified time points during the operation to evaluate the cardiovascular effects of spinal anesthesia in preeclamptic patients.
Renal Function Parameters Post-Spinal Anesthesia | Postoperative 4th hour
  Evaluation of postoperative serum creatinine levels to assess renal function in the early postoperative period.
Renal Function Parameters Post-Spinal Anesthesia | Postoperative 4th hour
  Evaluation of postoperative eGFR levels to assess renal function in the early postoperative period.

OTHER OUTCOMES:
Incidence of Spinal Anesthesia-Related Hypotension | Within the first 30 minutes after spinal anesthesia
  Number and percentage of patients who experience hypotension (defined as a >20% decrease from baseline systolic blood pressure) following spinal anesthesia.
Total Intraoperative Vasopressor Requirement | Intraoperative period
  otal dose of vasopressors (e.g., ephedrine or phenylephrine) administered to treat spinal-induced hypotension.

CONTACTS AND LOCATIONS:
Overall Officials: Nihan Aydın Güzey, Principal Investigator — Ankara City Hospital Bilkent
Locations (1):
- Ankara City Hospital, Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No